CLINICAL TRIAL: NCT03093987
Title: Critical Care Ultrasound Oriented Shock Treatment in ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, tongjuan ZOU, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: West China Hos
Record Dates: First submitted 2017-03-06; First posted 2017-03-28 (Actual); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Shock
Keywords: Shock; Critical Care Ultrasound; Lactate; Mortality; Prognosis
MeSH Terms: conditions — Shock

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): usual care
- critical care ultrasound (Experimental): Circulation management will be adjusted according to the results of critical ultrasound combined with clearance of lactic acid in patients with shock.
  Interventions: Other: Critical care ultrasound

INTERVENTIONS:
Other: Critical care ultrasound — Circulateory will be managed according to the result of critical ultrasound joint clearance of lactic acid in patients with shock
  Arms: critical care ultrasound

SUMMARY:
Objective

To investigate whether critical care ultrasound oriented shock management in shock patients in intensive care unit(ICU) can improve outcome.

Methods

Randomized controlled research. Patients were randomly allocated to two groups. In the critical care ultrasound oriented shock management group (CUSS group), treatment was oriented by the findings of critical care ultrasound in each shock phase, while in the control group the decisions about the monitoring and management were made by the clinical team. The goal of treatments in both groups were decreasing lactate by 20% or more per 2 hours for the Optimization phase in shock management, and no increase lactate level when removing the fluid in de-escalation phase. The primary outcome measure were hospital mortality and 28-day mortality, the secondary outcome measure were the length of ventilation and the length of ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* SBP <90 mm Hg or MAP <65 mm Hg or SBP decrease >40mmHg or need vasoactive drugs；
* Skin that is cold and clammy，capillary refill time >4.5s，urine output of<0.5ml/Kg.hr and lactate >2mmol/L；
* SHOCK presented within 6 hr.

Exclusion Criteria:

* <18 years old；
* Pregnancy；
* Patient or family member refuse to be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2017-10-28 (Actual); Study Completion 2017-10-28 (Actual)

PRIMARY OUTCOMES:
28-day mortality | through study completion,an average of 28 days
  28-day mortality

SECONDARY OUTCOMES:
the length of ICU stay | through study completion,an average of 28 days
  the length of ICU stay
the total length of hospital stay | through study completion,an average of 28 days
  the total length of hospital stay
the incidence of AKI | through study completion,an average of 28 days
  the incidence of AKI

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lichtenstein D. Fluid administration limited by lung sonography: the place of lung ultrasound in assessment of acute circulatory failure (the FALLS-protocol). Expert Rev Respir Med. 2012 Apr;6(2):155-62. doi: 10.1586/ers.12.13. PMID 22455488
- [Result] Schmidt GA, Koenig S, Mayo PH. Shock: ultrasound to guide diagnosis and therapy. Chest. 2012 Oct;142(4):1042-1048. doi: 10.1378/chest.12-1297. PMID 23032454
- [Result] Holm JH, Frederiksen CA, Juhl-Olsen P, Sloth E. Perioperative use of focus assessed transthoracic echocardiography (FATE). Anesth Analg. 2012 Nov;115(5):1029-32. doi: 10.1213/ANE.0b013e31826dd867. Epub 2012 Oct 9. No abstract available. PMID 23051882
- [Result] Lichtenstein DA, Meziere GA. Relevance of lung ultrasound in the diagnosis of acute respiratory failure: the BLUE protocol. Chest. 2008 Jul;134(1):117-25. doi: 10.1378/chest.07-2800. Epub 2008 Apr 10. PMID 18403664
- [Result] Manno E, Navarra M, Faccio L, Motevallian M, Bertolaccini L, Mfochive A, Pesce M, Evangelista A. Deep impact of ultrasound in the intensive care unit: the "ICU-sound" protocol. Anesthesiology. 2012 Oct;117(4):801-9. doi: 10.1097/ALN.0b013e318264c621. PMID 22990179
- [Result] Vincent JL, De Backer D. Circulatory shock. N Engl J Med. 2013 Oct 31;369(18):1726-34. doi: 10.1056/NEJMra1208943. No abstract available. PMID 24171518
- [Result] Bhat SR, Swenson KE, Francis MW, Wira CR. Lactate Clearance Predicts Survival Among Patients in the Emergency Department with Severe Sepsis. West J Emerg Med. 2015 Dec;16(7):1118-26. doi: 10.5811/westjem.2015.10.27577. Epub 2015 Dec 8. PMID 26759665